CLINICAL TRIAL: NCT06560970
Title: A Technology-based Psychosocial Intervention to Support Social Engagement and Well-being in Older Adults With HIV
Acronym: COPPEhR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-08026417; R21AG074832 (NIH)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: HIV Diagnosis
Keywords: Technology; Computer; Social Engagement; Well-being; Older Adults

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be blind to their assigned condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPPEhR Intervention (Experimental): Participants will have access to the COPPEhR system which will provide social support and engagement among older adults diagnosed with HIV.
  Interventions: Behavioral: COPPEhR Intervention
- Device-only Control Condition (Placebo Comparator): Participants will have access to a device only without the COPPEhR system.
  Interventions: Behavioral: Device-only Control Condition

INTERVENTIONS:
Behavioral: COPPEhR Intervention — Participants will receive access to the COPPEhR system which will provide social support and engagement among older adults diagnosed with HIV.
  Arms: COPPEhR Intervention
Behavioral: Device-only Control Condition — Participants will have access to a device only without the COPPEhR system.
  Arms: Device-only Control Condition

SUMMARY:
Older people with HIV (OPH) often live with significant mental health challenges such as social isolation, loneliness, and depression. The objectives of this study are to develop and test the usability and feasibility of a technology-based psychosocial intervention program designed to: enhance social engagement and support; facilitate resource access and education; reduce loneliness; and improve well-being among older adults with HIV who are long-term survivors (diagnosed with HIV ≥ 20 years). The program, Connecting Older Positive People to Enhance Health and Resilience (COPPEhR), will build on Dr. Sara Czaja's PRISM (A Personal Reminder and Information Management System for Seniors) platform, and will be an easy-to-use software application (app), preloaded onto a standard device, designed to support social connectivity, memory, and access to resources for older adults at risk for isolation and the programs and services available at the Center for Special Studies (CSS) at Weill Cornell Medicine (WCM). This protocol covers Phase 2 of the study, which will be a pilot randomized controlled efficacy trial will compare the COPPEhR intervention to a device-only control condition. Participants in the control condition will receive the same device as those in the COPPEhR condition without the COPPEhR application. The specific aims of this developmental project are to evaluate the feasibility, usefulness, and usability of a state-of-the art technology-based multicomponent COPPEhR intervention for aging adults with HIV. Our hypothesis is the COPPEhR intervention will be feasible, usable and useful. The hypothesis is that those that use the COPPEhR app will experience less loneliness, less depression, and less social isolation and more social support, more resilience, and more connectivity than those that do not use the COPPEhR app.

DETAILED DESCRIPTION:
The development of modern antiretroviral therapies has increased the life expectancy of people living with HIV (PLWH) allowing them to survive into older ages. Older people with HIV (OPH) have an enhanced risk of developing multiple chronic conditions, such as cardiovascular disease, kidney and liver disease, cancer, and cognitive impairment. Also, especially for those who had treatment early, HIV remains stigmatized. OPH live with significant mental health interdependent challenges such as social isolation, loneliness, and depression. Because of stigma and protective withdrawal behaviors, OPH also tend to have limited social networks and opportunities for engagement. In a recent study of people ≥ 50 years of age with HIV, 58% of the sample (N=356) reported experiencing loneliness. Moore and colleagues, found that older adults with HIV in their sample spent a considerable amount of time at home alone engaged in solitary activities.

The consequences of social isolation include lower quality of life and life satisfaction and poorer mental, physical, and cognitive health. With respect to OPH, studies have shown that loneliness is associated with substance abuse, depression, and poorer quality of life. So-Armah and colleagues, using data from the Veterans Aging Cohort study, found that depressive symptoms were associated with all-cause mortality among US veterans with HIV but not among those without HIV infection. To date, there has been limited intervention research directed at psychosocial issues among OPH, especially long-term survivors. In fact, a recent systematic review of psychosocial interventions for older adults with HIV/AIDS found a paucity of psychosocial interventions and few randomized trials and highlighted a need for home-based interventions to enhance the quality of life for adults aging with HIV. As noted by the National Institutes of Health Office of AIDS Research Working Group on HIV & Aging, research focused on social isolation and behavior is critical for this population.

Technology-based interventions provide a potential solution for enhancing access to instrumental and social support for older adults with HIV and offer unparalleled flexibility in information presentation and facilitates broad implementation of applications. As noted by a recent report from the National Academies of Science, Engineering, and Medicine that focused on social isolation, "technology provides an important set of opportunities for the 'toolkit' of strategies that can help prevent or mitigate social isolation and loneliness in older adults (pg. 9-38)." Studies have examined the impact of access to the Internet on well-being and social outcomes for older adults, and the results are encouraging. For example, use of the Internet was shown to decrease loneliness and increase social contact among a sample of higher use of social technology was linked to higher ratings of health and well-being and lower depressive symptoms. The links between use of social technology and these outcomes were mediated by reductions in loneliness. The investigators conducted an randomized control trial (RCT) that evaluated PRISM, a software system that supports social connectivity, memory, and information access, with older adults at risk for social isolation. Findings indicated that use of PRISM resulted in significantly less loneliness, increased social support and well-being, and an increase in device comfort and proficiency at 6 months.

Recent studies support the importance and acceptability of using technology for aging adults with HIV. Moore and colleagues8 found that older adults with HIV were able to use smart phones to collect ecological momentary assessment data. Findings from a recent study indicated that OPH that participated in an online mindfulness intervention showed reductions in depression, anxiety, and loneliness. The objectives of this proposed development study are to develop and evaluate a technology-based psychosocial intervention, Connecting Older Positive People to Enhance Health and Resilience (COPPEhR), designed to increase social and cognitive engagement and resource access, reduce loneliness, and improve well-being among OPH. COPPEhR will be delivered on a device via an app and the features will be guided by Activity Theory, models of Successful Aging, and Social Engagement, which underscore that social and cognitive engagement are integral to successful aging and that the benefits of social and meaningful engagement include better emotional, physical and cognitive health.

In accordance with these theories, the features of COPPEhR will provide opportunities for social support and connection, social network expansion (e.g., online support groups, buddies/interest groups) and expansion of social capital (community feature) which the investigators postulate will enhance social engagement, which will in turn be linked to less loneliness and better well- being (e.g., less depression) COPPEhR will also be based on our prior NIH funded work; services available at the Center for Special Studies (CSS), which has a clinic for OPH; the resources of the Center on Aging and Behavioral Research (CABR) (Czaja, Director); and the Center for Research and Education on Aging and Technology Enhancement (CREATE) (Czaja, PI).

ELIGIBILITY:
Inclusion Criteria:

1. Age 50+
2. HIV diagnosis for at least 15 years
3. Center for Special Studies (CSS) patient
4. Able to read English at 6th grade level
5. Visually able to read a device screen
6. Adequate cognitive status (score above 34) to interact with the technology assessed by the Telephone Interview for Cognitive Status - modified (TICS-M)
7. Plan to remain in the area for the next 9 months

Exclusion Criteria:

1. Not a Center for Special Studies (CSS) patient
2. Blind or have visual impairments that limit their ability to view the technology
3. Deaf or have hearing impairments that limit their ability to use the technology
4. Has a mobility or dexterity impairment that would interfere with the use of a device, mouse, or a keyboard (e.g., tremors, arthritis, etc.)
5. Severe psychosis (e.g., aggression)
6. Severe cognitive impairment that limits their ability to use the technology
7. Participants who do not meet the inclusion criteria.
8. Participants in previous COPPEhR usability testing

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Mean Difference of Perceived Usefulness and Perceived Ease of Use Questionnaire | Post-randomization at month 3 and month 6
  Utilizing a 12-item scale (Perceived Ease of Use Questionnaire) which includes two subscales (perceived usefulness and perceived ease of use) with Likert response scales ranging from 1 (Strongly disagree) - 7 (Strongly agree). The total score ranges from 12 - 84. The responses to the items are summed for each of the subscales. Higher scores indicate perceived ease of use of the COPPEhR program.
Mean Difference of System Evaluation Questionnaire | Post-randomization at month 3 and month 6
  The COPPEhR system or device evaluation will be assessed by evaluating participants' perception of the features of the system. Utilizing an 11-item scale with Likert response scales ranging from 1 (Strongly disagree) - 5 (Strongly agree). The total score ranges from 11 - 55. Higher scores indicate higher degrees of satisfaction with the COPPEhR system, training, technical support.

SECONDARY OUTCOMES:
Mean Difference in Score of reported depression, assessed using the Center for Epidemiological Studies-Depression (CES-D) Scale | Post-randomization at Baseline, month 3, and month 6
  The CES-D is a self-report depression scale for research in general population. It is a 20 item questionnaire consisting of likert response scales ranging from 0-3 points. The total score range is 0 - 60 points. Higher scores indicate participants have a greater level of self reported depression.
Change in Loneliness as Measured by UCLA Loneliness Scale | Post-randomization at Baseline, month 3, and month 6
  To measure degree of loneliness. The 3rd version of the UCLA Loneliness Scale includes positively worded or non-lonely items. It is a 20 item questionnaire consisting of likert response scales ranging from 0-3 points. Higher score indicates a greater degree of loneliness. Range (0-60)
Mean Difference in Score of Quality of Life, assessed using The Quality of Life Questionnaire | Post-randomization at Baseline, month 3, and month 6
  Will assess the participant's quality of life by having the participant rate different aspects of their life using one of four words: poor, fair, good, or excellent. They are instructed to think about different aspects of their life, like physical health, energy, family, money, and others to assess their situation in each area.
  The Quality of Life questionnaire is a 13-item scale with Likert response scales ranging between 1 and 4 points. The measure's total score can range between 13 - 52 points. A higher total score is reflective of a higher quality of life while a lower score is reflective of a poorer quality of life.
Mean Difference in score of participants self-reported health, assessed using the 36-Item Short Form Health Survey questionnaire (SF-36 Short Form) | Post-randomization at Baseline, month 3, and month 6
  The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. The total measure scores range from 0 - 100. Lower scores = more disability, higher scores = less disability. The 8 subscales or domains are as follows: Physical functioning (10 items); Role limitations due to physical health (4 items); Role limitations due to emotional problems (4 items); Energy/fatigue (4 items); Emotional well-being (5 items); Social functioning (2 items); Pain (2 items); General health (5 items).
Mean Difference in score of participants self-reported Resilience, assessed by BRS - Brief Resilience Scale | Post-randomization at Baseline, month 3, and month 6
  The BRS Brief Resilience Scale will assess a person's self-perceived ability to bounce back or recover from stress. This questionnaire/scale has six items. It uses a 5-point Likert scale with 5 response categories - Strongly Disagree, Somewhat Disagree, Neither Agree nor Disagree, Somewhat Agree and Strongly Agree. The total score ranges from 6 - 30. Higher scores indicates a greater level of resilience.
Mean Difference in Score of Social Support and Connectivity Assessed using The Social Connectedness Measure | Post-randomization at Baseline, month 3, and month 6
  Scales used to measure two aspects of social isolation: social disconnectedness and perceived isolation, as well as perceived availability of social support. The Social Connectedness measure is a 15-item scale consisting of 3 sections with different likert response scale. Section 1 is a 4 item scale ranging from 0 - 5 points (20 total points). Section 2 is a 6-item scale ranging from 1 - 3 points (18 total points). Section 3 is a 5-item scale ranging from 1 - 5 points (25 total points). The total score ranges from 11 - 63. A higher total score is reflective of increased connectedness, with items 5-7 and items 11-15 reverse scored. Total scores will be summed and then a mean difference in score will be calculated.
Social Engagement using the Lubben Social Network Index (LSNS-6) | Post-randomization at Baseline, month 3, and month 6
  The Lubben Social Network Index (LSNS-6) will assess social engagement including family and friends. This scale has 6 items. The score is computed by adding the response of all items. The score ranges between 0-30 with higher scores indicating more social engagement.
Medical Outcome Study: Social Support Survey Instrument | Post-randomization at Baseline, month 3, and month 6
  This is a 19-item questionnaire that measures emotional/informational support, tangible support, affectionate support, positive social interaction, and one additional miscellaneous item. The survey/instrument consists of four separate social support subscales and an overall functional support index. The total score ranges from 19 - 95. A higher score for an individual scale or for the overall support index indicates more support.
Mean Difference in score of Social Isolation using the Friendship Scale | Post-randomization at Baseline, month 3, and month 6
  This questionnaire/scale has a total of 6 items measuring perceived social isolation. The time frame of the questions is set at 4 weeks. The scale used for this questionnaire is as follows: Almost always = "0"; Most of the time = "1"; About half the time = "2'; Occasionally = "3"; and Not at all = "4". The score range is 0-24. A high score represents social connectedness and a score of "0" indicates complete social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Czaja, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan for resource sharing is based on the National Institutes of Health/National Institute on Aging (NIH/NIA) Data Sharing Policy. The investigators plan, consistent with the NIH goals of data sharing, is to promote use of the rich COPPEhR database by the larger research community as this will further the impact of COPPEhR and expand possibilities for collaboration. It will also allow other researchers to expedite the translation of the research findings into knowledge, products, and procedures. Further, the plan is devised to make the data as widely and freely available as possible while at the same time safeguarding the privacy of participants and protecting confidential and proprietary data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data from research projects will be made available no later than acceptance of publication of the main findings from the final data set. There is no end date to access the data from the research projects.
Access Criteria: The investigators agree to share the data with researchers working under an institution with Federal Wide Assurance who agree to a data sharing agreement that stipulates protection of participant privacy and data confidentiality, acknowledgement of COPPEhR, that the data will be used for research purposes only, and that the data will not be transferred to other users. The computerized data will include raw data, derived variables, all necessary documentation as described in the National Archive of Computerized Data on Aging depositor agreement. All data will be de-identified. The investigators will follow the guides published by the US Department of Health and Human Services in this respect. Each data set will include data documentation to ensure that others can use the data set and to minimize confusion. Information about where and how to locate and access the data will be available in any publications and presentations authored by COPPEhR investigators.